CLINICAL TRIAL: NCT01199978
Title: Hearing Outcomes Using Fractionated Proton Radiation Therapy for Vestibular Schwannoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-218
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Vestibular Schwannoma; Acoustic Neuroma
Keywords: radiation; fractionated proton radiation
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fractionated Proton Radiation (Other): Single arm study, delivering fractionated radiation with a technique (proton therapy) that may be associated with reduced side effects
  Interventions: Radiation: Fractionated proton radiation; Drug: Losartan

INTERVENTIONS:
Radiation: Fractionated proton radiation — Given daily for approximately 5.5 weeks
Drug: Losartan — 25mg or 50mg daily, oral administration, for approximately 6 months.
  Other Names: Cozaar

SUMMARY:
In this research study we are looking at another type of radiation called proton radiation which is known to spare surrounding normal tissues from radiation. The proton radiation will be delivered using fractionated stereotactic radiotherapy (FSRT) to improve localization of the small tumor target. Proton radiation delivers minimal radiation beyond the area of the tumor. This may reduce side effects that patients would normally experience with conventional radiation therapy. In this research study, we are looking to determine the effects of fractionated proton radiotherapy on long-term hearing preservation and controlling tumor growth.

DETAILED DESCRIPTION:
* Proton radiation will be delivered daily for approximately 5.5 weeks. Participants will be assessed weekly for any side effects they may be experiencing.
* Participants will have a follow-up visit 6 months after their last proton radiation treatment and then every year from the time of treatment completion for 5 years. The following tests and procedures will be performed at these visits: medical history, physical exam, MRI scan, comprehensive hearing tests and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* MRI confirmed unilateral vestibular schwannoma within 8 weeks prior to study entry
* Measurable disease, defined as a lesion that can be accurately measured in at least one dimension
* No prior radiotherapy with dose delivered to structures in proximity to the internal acoustic canal is allowable
* Participants must have baseline "useful hearing" defined at the discretion of the treating physician in the irradiated ear
* 18 years of age or older
* Life expectancy of greater than 60 months
* Karnofsky performance status 60 or greater
* Diagnosis of neurofibromatosis 2 (NF2) is permitted
* Women of child-bearing potential and men must agree to use adequate contraception during the interval of irradiation
* Able to tolerate the supine position as required for the radiation treatment unit and able to tolerate rotation needed for treatment delivery
* Able to tolerate the standard immobilization device that typically utilizes a dental impression mouth piece and thus requires breathing through the nasal passage.
* Willing and able to comply with comprehensive audiologic testing, at baseline prior to radiation therapy, at 6 months from treatment completion, and at annual timepoints for 5 years after completion
* Baseline Systolic Blood Pressure (BP) > 100mm Hg. This is based on the average of two values - separate seated, resting measurements taken five minutes apart. BP does not need to be checked in both arms unless a reading is below 110 mm Hg, in which case the other arm can be checked as well. If BP is checked in both arms, the higher value is deemed accurate for calculating the average.

Exclusion Criteria:

* Participants who have had prior radiotherapy, with dose delivered to structures in proximity to the internal acoustic canal (IAC).
* Participants with tumors (or residual tumor after surgery) measuring > 3cm in greatest dimension
* Participants may not be receiving any other study agents
* History of adverse reaction to radiotherapy
* Participants may not already be on losartan, other angiotensin II type I receptor blocker (ARB), or on an angiotensin-converting enzyme (ACE) inhibitor prior to enrollment of this study.
* Participants receiving any medications or substances that are known to cause ototoxicity are ineligible
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Individuals with a history of malignancy are ineligible except for the following circumstances. Individuals with a history of malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be a low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy
* Patients with co-existing major ear disease, such as chronic otitis, Menieres disease, or otosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Characterization of long-term hearing effects | 5 years
  Characterization of long-term hearing effects of fractionated proton therapy in patients with vestibular schwannomas.

SECONDARY OUTCOMES:
Local control rate after fractionated proton radiation | 5 years
Delineation of dosimetric parameters after fractionated proton radiation | 5 years
  The distribution of dosimetric parameters will be summarized, and their correlation to clinical outcomes, including hearing loss, will be explored.
Incidence of second tumors after fractionated proton radiation | 5 years
Toxicity profile of Losartan given concurrently with proton radiation | 5 years
  Toxicities associated with losartan before, during and after proton radiation will be summarized by grade according to CTCAE 4.0. The losartan cohort of 10 participants will provide 90% confidence interval of maximal width +/-27% based on the exact binomial distribution.
Impact of Losartan on hearing preservation | 5 years
Impact of Losartan on circulating biomarkers | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Helen A. Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Saraf A, Pike LRG, Franck KH, Horick NK, Yeap BY, Fullerton BC, Wang IS, Abazeed ME, McKenna MJ, Mehan WA, Plotkin SR, Loeffler JS, Shih HA. Fractionated Proton Radiation Therapy and Hearing Preservation for Vestibular Schwannoma: Preliminary Analysis of a Prospective Phase 2 Clinical Trial. Neurosurgery. 2022 May 1;90(5):506-514. doi: 10.1227/neu.0000000000001869. PMID 35229827